CLINICAL TRIAL: NCT00346411
Title: Health Outcomes in Rheumatoid Arthritis
Acronym: HORA
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00001359
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; mood; adherence; medication
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This research is being done to help us learn about how different factors related to treatment affect rheumatoid arthritis (RA). This is not a treatment study. We will follow the patient for one year as he or she receives usual treatment from his or her rheumatologist. Up to 360 adults with RA may join this study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 19 or older
* Current active, adult-onset rheumatoid arthritis who meet American College of Rheumatology (ACR) criteria for RA and have: (ACR functional class I-III), defined as:
* 3 or more swollen or tender joints and
* Morning stiffness of 45min or longer
* OR judged by their rheumatologist to have active disease
* No evidence of other inflammatory diseases (e.g., Crohn's, IBS)
* Functional class I, II or III

Exclusion Criteria:

* Individuals with significant cardiovascular disease (CHF, stroke, MI)
* Unwilling to have medications monitored and/or comply with protocol
* Not fluent in English
* Planning to move from area within next year or change health insurance (which would preclude ongoing care by a Johns Hopkins rheumatologist)
* Enrolled in study evaluating efficacy of new or existing RA medications

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with rheumatoid arthritis and receiving treatment for this condition from a rheumatologist
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2005-09-01 (Actual); Primary Completion 2011-12-12 (Actual); Study Completion 2011-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Bartlett, PhD, Principal Investigator — Johns Hopkins School of Medicine; Cynthia S Rand, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Campus, Baltimore, Maryland, United States